CLINICAL TRIAL: NCT05909254
Title: Application of Surgical Templates in the Surgical Exposure of Impacted Canines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, senior lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEDCD54
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Impacted Tooth
Keywords: surgical exposure; open eruption technique
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palatally impacted canine exposure using a surgical template (Experimental)
  Interventions: Other: Palatally impacted canine exposure using a surgical guide
- Palatally impacted canine exposure using the conventional free-hand method (Experimental)
  Interventions: Other: Palatally impacted canine exposure using the conventional free.hand method

INTERVENTIONS:
Other: Palatally impacted canine exposure using a surgical guide — Under local anaesthesia the tissues covering the palatally impacted canine are removed with the help of a surgical guide to expose the tooth, to allow the bonding of an attachment on its surface for orthodontic traction.
  Arms: Palatally impacted canine exposure using a surgical template
Other: Palatally impacted canine exposure using the conventional free.hand method — Under local anaesthesia the tissues covering the palatally impacted canine are removed to expose the tooth, to allow the bonding of an attachment on its surface for orthodontic traction. The surgeon relies on the surgical plan and their experience to localize the impacted canine.
  Arms: Palatally impacted canine exposure using the conventional free-hand method

SUMMARY:
The first choice therapy in case of palatally impacted canines is their exposure and orthodontic eruption to improve facial esthetics and prevent pathologies associated with impacted teeth and Temporomandibular Joint Disorders. Current solutions in digital dentistry allow the registration of three dimensional imaging datasets such as cone beam computed tomography (CBCT) and digital impression of the dentition and soft tissues obtained via intraoral scanning using orthodontic planning software. This allows the surgeon to visualize the position of the impacted canine prior to surgery and to design and manufacture a surgical guide to aid in the localization of the impacted tooth during surgery.

The aim of this randomized clinical trial is to assess the feasibility of surgical exposure of palatally impacted upper canines with open-eruption technique using a surgical template. The secondary purpose of this study is to compare this method with the conventional free-hand surgical exposure.

Patients included in this study are randomly assigned to two study groups. In Group 1 surgical exposure for open eruption of palatally impacted canines is performed following virtual planning using a surgical template. In Group 2 surgical exposure for open-eruption of palatally impacted canines is carried out using the conventional free-hand method.

We hypothesize that guided exposure of the impacted canines will be as successful as the conventional method with shorter surgical intervention and higher associated costs.

DETAILED DESCRIPTION:
Objectives The aim of this randomized clinical trial is to assess the feasibility of surgical exposure of palatally impacted upper canines with open-eruption technique using a surgical template. The secondary purpose of this study is to compare this method with the conventional free-hand surgical exposure. Our null-hypothesis is that there will be no significant differences in the outcome measures between the two methods.

Materials and methods

Groups

* Group 1 (test group): Surgical exposure for open eruption of palatally impacted canines following virtual planning using a surgical template.
* Group 2 (control group): Surgical exposure for open-eruption of palatally impacted canines using the conventional free-hand method.

Simple randomization is performed to determine whether patients are included in the test or control group. 20 patients are recruited per group. During continuous recruiting, sample size calculation is to be carried out to determine the actual number of patients included in this study.

Surgical planning The upper jaw of the patient is scanned using an intraoral scanner (IOS, Trios 4, 3Shape, Copenhagen, Denmark). Cone beam tomography (CBCT) scans (Green X, Vatech, Hwaseong, Korea) are performed before surgical exposure to assess the position, angulation, possible dilaceration, and bone coverage of the impacted canines. The scanning conditions are constant at 200 μm isotropic voxel size with 360◦ rotation, 94 kiloVolt (kV) tube voltage, 7.2 miliAmper (mA) tube current, and 9 s exposure time with a field of view of 15 × 8 cm. In the test group OnyxCeph³™ software is used to register the standard tessellation language (STL) file of the digital impression with the Digital Imaging and Communications in Medicine (DICOM) data of the pre-operative CBCT reconstruction by surface registration. A surgical template is designed to cover the palate, incisal, and occlusal surfaces of the dentition with an opening that outlines the window to be prepared to expose the impacted canine. Fused deposition modeling (FDM) is used for the rapid prototyping of the surgical template (FlashForge Creator Pro 4, Zhejiang Flashforge 3D Technology Co., Ltd, Jinhua City, China) using polylactic acid filament (PLA).

Surgery In both groups patients rinse their oral cavity with 0.2% chlorhexidine solution for 1 min before surgery and surgical interventions are performed under local anesthesia. In the test group the fit of the surgical template is a checked and a surgical laser (SiroLaser Blue, Dentsply Sirona, Charlotte, North Carolina, U.S.A.) is used for the exposure of the impacted canine. In the control group the surgeon relies on the surgical plan and their experience to localize the impacted canine. The attachment is bonded to the exposed canine by an orthodontist. Patients are instructed to clean the wound using toothpaste and toothbrush and to rinse with 0.2% chlorhexidine solution in the morning and in the evening for a week starting on the day after surgery. Anti-inflammatory drugs (25 mg diclofenac three times a day for 3 days) are prescribed to control postoperative pain

Management of participant-bias Surgical planning and interventions are performed by a skilled surgeon. The clinician performing the exposure of the impacted canine is not involved in the evaluation of the outcome measures. The examiner carrying out the measurement of the outcome variables was blinded to the surgical modality used during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 11-18 of the Department of Community Dentistry, Semmelweis University, who need surgical exposure and orthodontic eruption of their palatally impacted canines on one or both sides during their orthodontic treatment are included in this study.

Exclusion Criteria:

* Uncontrolled systemic diseases that contraindicate orthodontic treatment or minor dental surgery,
* Trauma in the patient's history in the vicinity of the surgical site.
* Dental abnormalities (hyperdontia, hypodontia, etc.),
* Congenital craniofacial disorders,
* Permanent teeth extraction-based treatment,
* Periodontal disease,
* Cases in which the canine is to be brought into the position of the lateral incisor,
* Agenesis of lateral incisors on the impaction side,
* Documented learning disability,
* Insufficient oral hygiene, and
* Non-compliance during the combined orthodontic-surgical treatment.
* Smoking

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Success of the intervention | on the day of the surgery
  Measures if an attachment could be bonded to the impacted tooth during the surgery.
Success of the open eruption technique | 1 year
  Measures whether the canine erupts in its correct place in the dentition following tha application of orthodontic forces.

SECONDARY OUTCOMES:
Surplus costs of surgical planning and manufacturing the surgical guide | through study completion, an average of 1 years
  Measures the excess costs of the design and manufacture of surgical guides used in Euro.
Duration of the surgical intervention | during surgery
  Measures the duration of the surgery in minutes.
Postoperative pain | 1 week
  Pain and recovery reported by the patient after surgery, measured on 100 mm visual analog scale (VAS) on the evening of the intervention and in the following 7 days. 0 is the lowest score, which means that the patient experienced no pain at all following surgery, 100 is the highest score refering to the worst pain the patient had ever experienced previously.
Intra- and postoperative complications associated with surgery | through study completion, an average of 1 years
  Number of cases where bleeding, damage to neighboring teeth, roots, and anatomical structures, nerve damage, antro-oral communication or fistula, inflammation is observed during follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Community Dentistry, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kivovics M, Szanyi SM, Takacs A, Repasi M, Nemeth O, Mijiritsky E. Computer-assisted open exposure of palatally impacted canines for orthodontic eruption: A randomized clinical trial. J Dent. 2024 Aug;147:105110. doi: 10.1016/j.jdent.2024.105110. Epub 2024 Jun 20. PMID 38906453